CLINICAL TRIAL: NCT03275844
Title: Physical Capacity and Activity in Children With Congenital Heart Disease in Chile
Brief Title: Physical Capacity and Activity in Children With Congenital Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rodrigo Torres (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Torres, Assistant Professor, University of Chile
Organization: University of Chile (Other)
Other Study IDs: 2017-01
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Heart Defects, Congenital; Tetralogy of Fallot
Keywords: Physical activity; Physical capacity; Children
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Children with congenital heart disease
  Interventions: Procedure: Physical activity assessment
- Group 2: Control healthy subjects
  Interventions: Procedure: Physical activity assessment

INTERVENTIONS:
Procedure: Physical activity assessment — Assessment of Moderate-to-vigorous physical activity

SUMMARY:
Congenital malformations correspond to defects in organ morphogenesis identifiable at birth or intrauterine life, affecting 2-3% of births. Inside of these malformations, Congenital Heart Disease corresponds, in particular, to structural defects of the heart or major blood vessels thereof may or may not be associated with other types of syndromes.The resolution is usually surgical.

Also, these patients present a decrease in physical fitness, psychological imbalance, lower quality of life and risk significant morbidity and mortality from respiratory infections among other problems.

This can have severe consequences for health in the medium and long term. The habits acquired during childhood and adolescence are determinant for the adult life, being relevant levels of activity and physical condition, especially in children with pathologies.

In this way, it is vital to know from childhood parameters that indicate the baseline state of these patients according to the levels of physical activity, exercise capacity, nutritional status and quality of life. These will be key indicators to take into account in the future, to adapt rehabilitation plans that will reduce the effects of their condition.

The objective of this protocol is To characterize the levels of Activity, and Physical Capacity of children with congenital heart disease regularly treated at the Cardiovascular Center of Dr. Luis Hospital Calvo Mackenna, compared to healthy children matched by age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Children with Tetralogy of Fallot corrected
* Age from 6 to 15 years
* Assistants to periodic control at HLCM Cardiovascular Center

Exclusion Criteria:

* Morbid obesity
* Musculoskeletal disorders that impede physical activity
* Neurological comorbidity
* Respiratory comorbidity in the last 30 days.
* Pacemaker users

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with congenital heart diseases
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity | 1 week
  Time in minutes of Moderate-to-vigorous physical activity

SECONDARY OUTCOMES:
Six minute walking test | 1 hour
  Walked distance in six minute walking test
Steps | 1 week
  mean of number of steps per day

CONTACTS AND LOCATIONS:
Overall Officials: Homero Puppo, MSc, Study Chair — Univeridad de Chile

IPD SHARING:
Plan to Share IPD: Undecided
Probably, All information will be public